CLINICAL TRIAL: NCT01102712
Title: Evaluation Study of Unilateral Bronchoscopic Thermal Vapor Ablation (BTVA) in Patients With Heterogeneous Emphysema and Upper Lobe Predominance
Brief Title: Bronchoscopic Thermal Vapor Ablation (BTVA) for Lung Volume Reduction
Acronym: BTVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptake Medical Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vapor-OUS
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: Emphysema; COPD; Lung Volume Reduction; BTVA
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTVA (Experimental)
  Interventions: Device: BTVA System

INTERVENTIONS:
Device: BTVA System — Unilateral Bronchoscopic Thermal Vapor Ablation for Lung Volume Reduction

SUMMARY:
To establish and confirm the safety and clinical utility of BTVA applied unilaterally for lung volume reduction in patients with upper lobe predominate heterogeneous severe emphysema.

DETAILED DESCRIPTION:
All subjects meeting the eligibility criteria and who provide written informed consent will be enrolled. Up to 3 segments in either the right or left upper lobe will be treated with a vapor dose of 10 calories per gram of lung tissue (10 cal/g). Targeted lobe for treatment will be based on lobar disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 40 and ≤ 75 years old
2. Diagnosis of heterogeneous emphysema with upper lobe predominance
3. FEV1 < 45% predicted
4. TLC > 100% predicted
5. RV > 150% predicted
6. 6-minute walk test > 140 meters
7. mMRC ≥ 2 (mMRC)
8. Non-smoking for 3 months
9. Optimized medical management and completed pulmonary rehabilitation

Exclusion Criteria:

1. Known α-1-antitrypsin deficiency
2. BMI < 15 kg/m2 or > 35 kg / m2
3. History of pneumothorax within previous 18 months
4. History of heart and / or lung transplant, lung volume reduction surgery (LVRS), median sternotomy, bullectomy, and/or lobectomy
5. Respiratory infections or recurring COPD exacerbations > 3 hospitalizations in past 12 months or active infection
6. History of the (EF) ≤ 40%; Stroke; Unstable Myocardial Ischemia; FEV1 < 15% predicted; DLCO < 20% predicted; pulmonary hypertension; indwelling pacemaker or implantable cardiac defibrillator (ICD); pregnancy or breastfeeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
increase in FEV1 ≥ 12% or a decrease in total St. George's Respiratory Questionnaire (SGRQ) score ≥ 4 points | 6 months

SECONDARY OUTCOMES:
Lobar volume reduction as determined by computed tomography (CT) analysis | 3 months
Changes in pulmonary function therapy | 3 months
Improvement in 6 minute walk distance | 3 months

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - Prince Charles Hospital, Chermside, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - LKH Klagenfurt, Klagenfurt
  - Otto-Wagner Hospital, Vienna
- Germany (5):
  - Zentralklinik Bad Berka, Bad Berka
  - Charite Campus Mitte, Berlin
  - Thoraxklinik Heidelberg, Heildelberg
  - Abteilung fur Pneumologie, Hemer
  - Klinikum Nurnberg, Nuremberg
- Mater Misericordiae University Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Herth FJ, Ernst A, Baker KM, Egan JJ, Gotfried MH, Hopkins P, Stanzel F, Valipour A, Wagner M, Witt C, Kesten S, Snell G. Characterization of outcomes 1 year after endoscopic thermal vapor ablation for patients with heterogeneous emphysema. Int J Chron Obstruct Pulmon Dis. 2012;7:397-405. doi: 10.2147/COPD.S31082. Epub 2012 Jul 18. PMID 22927751
- [Derived] Snell G, Herth FJ, Hopkins P, Baker KM, Witt C, Gotfried MH, Valipour A, Wagner M, Stanzel F, Egan JJ, Kesten S, Ernst A. Bronchoscopic thermal vapour ablation therapy in the management of heterogeneous emphysema. Eur Respir J. 2012 Jun;39(6):1326-33. doi: 10.1183/09031936.00092411. Epub 2011 Nov 10. PMID 22075481